CLINICAL TRIAL: NCT03578172
Title: Randomized, Controlled Trial to Assess the Efficacy of Human Menopausal Gonadotrophin Stimulation and Hormone Replacement Therapy for Endometrial Preparation Prior to Blastocyst Transfer in Moderate to Severe Intrauterine Adhesion Patients
Brief Title: HMG Stimulation Versus HRT for Endometrial Preparation Prior to Blastocyst Transfer in Moderate to Severe IUA Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYXM-2018001
Record Dates: First submitted 2018-06-24; First posted 2018-07-06 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Infertility, Female; Intrauterine Adhesion
MeSH Terms: conditions — Infertility, Female; Gynatresia | interventions — Menotropins; Hormone Replacement Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental-HMG stimulation group (Experimental): Women will be subjected to ovarian stimulation for endometrial preparation using human menopausal gonadotrophin before blastocyst transfer
  Interventions: Drug: human menopausal gonadotrophin
- Control-HRT group (Active Comparator): Women will be subjected to hormone replacement therapy for endometrial preparation before blastocyst transfer
  Interventions: Drug: hormone replacement therapy

INTERVENTIONS:
Drug: human menopausal gonadotrophin — experimental group:Women will be given HMG 37.5-150IU daily followed by monitoring of the follicular growth (folliculometry) when serum Estradiol (E2)<100pg/ml，progesterone (P)<1ng/ml. Final oocyte maturation will be induced by administration of human chorionic gonadotropin (HCG) when there will be at least one leading follicle ≥20mm in diameter followed by luteal phase support (using progesterone supplements) after 24 hours.
  Arms: Experimental-HMG stimulation group
Drug: hormone replacement therapy — Women will be given 17 β-estradiol hemihydrate 2 mg and estrogen gel 5 g daily from day 3 of the cycle then the endometrial thickness will be assessed on day 7 by transvaginal sonography (TVS). If the endometrium is ≥ 9 mm, luteal phase support (using progesterone supplements) will be started but if the endometrium is < 9 mm, estradiol will be continued until reaching appropriate endometrial thickness and then the luteal phase support will be started. The cycle will be cancelled If the estradiol administration >60 days.
  Arms: Control-HRT group

SUMMARY:
Evaluation of endometrial preparation using either human menopausal gonadotrophin (HMG) stimulation and hormone replacement therapy (HRT) prior to blastocyst transfer in patients with moderate to severe intrauterine adhesion (IUA).

ELIGIBILITY:
Inclusion Criteria:

* BMI 18~23 kg/m2
* Women with moderate to severe IUA as defined by the American Fertility Society classification (1988)
* Presence of at least 3 cryopreserved cleavage-stage embryos (including 1 good quality) or blastocysts

Exclusion Criteria:

* Using embryos from donor oocytes
* Preimplantation genetic diagnosis(PGD)/Preimplantation genetic screening(PGS) cycles
* Moderate or severe endometriosis
* Untreated unilateral or bilateral hydrosalpinx
* Uterine adenomyosis, uterine myoma (submucous,intramural myoma >4 cm),>1cm septate uterus, double uterus, bicornuate uterus, unicornuate uterus

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 10th week after embryo transfer
  Ongoing pregnancy is defined as the presence of a gestational sac with foetal heartbeat by transvaginal ultrasound at 10th week after embryo transfer（ET）

SECONDARY OUTCOMES:
Cycle cancellation rate | the day of embryo transfer
Implantation rate | 4th weeks after embryo transfer
  Sacs seen in early ultrasound divided by the number of embryos transferred
Clinical pregnancy rate | 4th weeks after embryo transfer
  Number of patients with ultrasound evidence of pregnancy divided by the number of embryo transfers
Early miscarriage rate | 12th weeks gestational age
  Number of losses of clinical pregnancies divided by number of clinical pregnancies
Biochemical pregnancy rate | 4th weeks after embryo transfer
  number of pregnancies with a transient elevation of serum human chorionic gonadotropin(β-hCG) level (>10 mIU/ml) divided by number of embryo transfers

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China